CLINICAL TRIAL: NCT02514044
Title: Transcranial Direct Current Stimulation and Melodic Intonation Therapy Combined With Dextroamphetamine in Chronic Stroke Patients With Non-fluent Aphasia; Safety and Efficacy Phase
Brief Title: Dextroamphetamine and tDCS to Improve the Fluency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Gerard Francisco, Chairman and Clinical Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-14-0354
Record Dates: First submitted 2015-06-04; First posted 2015-08-03 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Dextroamphetamine; Adderall; Speech Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Dexedrine+sham tDCS+speech therapy (Experimental): 10 mg Dexedrine and speech therapy for 10 days
  Interventions: Drug: Dexedrine; Behavioral: Speech Therapy; Device: Sham tDCS
- active tDCS+placebo+speech therapy (Experimental): 1.5 mA anodal tDCS and speech therapy for 10 days
  Interventions: Device: Active tDCS; Behavioral: Speech Therapy; Drug: Placebo
- Dexedrine+tDCS+speech therapy (Experimental): 10 mg Dexedrine, 1.5 mA anodal tDCS, and speech therapy for 10 days
  Interventions: Drug: Dexedrine; Device: Active tDCS; Behavioral: Speech Therapy
- sham stimulation+placebo+speech therapy (Experimental): Sham stimulation, placebo and speech therapy for 10 days
  Interventions: Behavioral: Speech Therapy; Drug: Placebo; Device: Sham tDCS
- Dexedrine+tDCS+Speech Therapy (Experimental): 10 mg Dexedrine, 1.5 mA anodal tDCS, and speech therapy for 1 day
  Interventions: Drug: Dexedrine; Device: Active tDCS; Behavioral: Speech Therapy
- placebo+tDCS+Speech Therapy (Experimental): 1.5 mA anodal tDCS, and speech therapy for 1 day
  Interventions: Device: Active tDCS; Behavioral: Speech Therapy; Drug: Placebo

INTERVENTIONS:
Drug: Dexedrine — 10 mg immediate release of Dexedrine
  Other Names: Adderall, Dexedrine
  Arms: Dexedrine+sham tDCS+speech therapy; Dexedrine+tDCS+Speech Therapy; Dexedrine+tDCS+speech therapy
Device: Active tDCS — 1.5 mA tDCS anodal tDCS
  Arms: Dexedrine+tDCS+Speech Therapy; Dexedrine+tDCS+speech therapy; active tDCS+placebo+speech therapy; placebo+tDCS+Speech Therapy
Behavioral: Speech Therapy — 60 min of speech therapy
  Other Names: Melodic Intonation Therapy
Drug: Placebo
  Arms: active tDCS+placebo+speech therapy; placebo+tDCS+Speech Therapy; sham stimulation+placebo+speech therapy
Device: Sham tDCS
  Arms: Dexedrine+sham tDCS+speech therapy; sham stimulation+placebo+speech therapy

SUMMARY:
The proposed study aims to evaluate safety and efficacy of combined dextroamphetamine (Dexedrine) and transcranial direct current stimulation (tDCS) with melodic intonation therapy (MIT) for treatment of aphasia after stroke. The target population is patients with chronic speech deficits due to a left hemisphere non-hemorrhagic stroke. Findings from this proposed project will help in the design of future larger studies.The safety phase will use cross-over, placebo controlled and single-blinded design. 10 participants with post stroke chronic non-fluent aphasia will undergo two experiments. To study the safety and effect of combined dextroamphetamine, tDCS and MIT therapy the study will use a parallel-groups, randomized, sham and placebo controlled, and double-blinded design in which 48 participants with post stroke chronic non-fluent aphasia will be randomly assigned to receive either 1) dextroamphetamine therapy with active stimulation, 2) placebo medication with active stimulation, 3) dextroamphetamine therapy with sham stimulation or 4) placebo medication with sham stimulation for the same duration.

DETAILED DESCRIPTION:
Two phases were planned for this study, as described below. The safety phase of the study was completed; however, due to limited funding, the efficacy phase was never started (that is, the efficacy phase was terminated).

SAFETY PHASE: The safety phase will use cross-over, placebo controlled and single-blinded design. 10 participants with post stroke chronic non-fluent aphasia will undergo two experiments. In the experiment 1, the subjects will receive 10 mg dextroamphetamine, 1.5 mA anodal tDCS to right inferior frontal gyrus (right Broca's area), and melodic intonation therapy. The two experiments of one time intervention will be separated by 1 week of washout and when the subjects come back for experiment 2, any later side effects will be evaluated. In the experiment 2, the subjects will receive placebo medication with anodal tDCS to right IFG (Broca's area) and melodic intonation therapy. During the experiments, thirty minutes before stimulation, participants in the active drug experiment (n=10) will take 10 mg dextroamphetamine per oral -experiment 1- and participants in the placebo drug experiment will take placebo pill per oral -experiment 2-. During the 20 minute stimulation phase, the participants (n=10) will receive anodal tDCS (1.5 mA) on ipsilesional right inferior frontal gyrus (Broca's area). All participants will simultaneously receive melodic intonation therapy for duration of an hour during and after 20 minutes of stimulation.

EFFICACY PHASE: To study the safety and effect of combined dextroamphetamine, tDCS and MIT therapy the study will use a parallel-groups, randomized, sham and placebo controlled, and double-blinded design in which 48 participants with post stroke chronic non-fluent aphasia will be randomly assigned to receive either 1) dextroamphetamine therapy with active stimulation, 2) placebo medication with active stimulation, 3) dextroamphetamine therapy with sham stimulation or 4) placebo medication with sham stimulation for the same duration. The subjects from the previous step of the study will be asked to participate to this step. Thirty minutes before stimulation participants in the active drug groups, group 1 (n=12) and group 3 (n=12) will take dextroamphetamine 10 mg per oral and participants in the placebo groups, group 2 (n=12) and group 4 (n=12) will take placebo pill per oral. During the 20 minute stimulation phase, the participants in the active stimulation groups, groups 1 (n=12) and 2 (n=12) will receive anodal tDCS (1.5 mA) on right inferior frontal gyrus (Broca's area), and participants in the sham control groups, group 3 (n=12) and group 4 (n=12) will receive sham stimulation. All participants will simultaneously receive melodic intonation therapy for duration of an hour during and after 20 minutes of stimulation. Treatment will be administered at an intensity of 5 sessions per week for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* Native English proficiency;
* Nonfluent speech;
* Premorbid right handedness;
* Non-hemorrhagic left hemispheric stroke at least 6 months prior to the investigation.
* No contraindications for MRI (only subjects who will undergo MRI scan).

Exclusion Criteria:

* Hypersensitivity or idiosyncrasy to dextroamphetamine or to other sympathomimetic agents;
* Pregnant or trying to become pregnant;
* Active alcohol abuse, illicit drug use or drug abuse or significant mental illness;
* Subjects receiving alpha adrenergic antagonists or agonists;
* Any history of epilepsy;
* Any condition that would prevent the subject from giving voluntary informed consent;
* An implanted brain stimulator;
* Aneurysm clip or other metal in the brain;
* Enrolled or plans to enroll in an interventional trial during this study;
* Scalp wounds or infections;
* Previous stroke with residual deficits (TIAs not a reason for exclusion);
* A concurrent progressive neurologic disorder, acute coronary syndrome, severe heart disease (NYHA Classification > 3), or other major medical condition;
* Advanced atherosclerosis, Unstable cardiac dysrhythmia or uncontrolled hypertension (>160/100 mm Hg), or untreated hyperthyroidism;
* Diagnosis of glaucoma
* During or within 14 days following the administration of monoamine oxidase inhibitors;
* Subjects requiring palliative care;
* Terminal medical condition such as AIDS or cancer;
* Subjects unable to comprehend or follow verbal commands;
* Based on PI's or local physician's assessment patient unable to tolerate the trial procedure due to medical condition;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard E Francisco, MD, Principal Investigator — University of Texas Health Science Center at Houston, Department of Physical Medicine and Rehabilitation
Locations (1):
- University of Texas Health Science Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexedrine+tDCS+Speech Therapy, Then Placebo+tDCS+Speech Therap: 10 mg Dexedrine, 1.5 mA anodal tDCS, and speech therapy for 1 day Dexedrine: 10 mg immediate release of Dexedrine Active tDCS: 1.5 mA tDCS anodal tDCS Speech Therapy: 60 min of speech therapy
  Placebo, 1.5 mA anodal tDCS, and speech therapy for 1 day Active tDCS: 1.5 mA tDCS anodal tDCS Speech Therapy: 60 min of speech therapy Placebo
Period: Dexedrine+tDCS+Speech Therapy (1 Day)
Arm/Group | Dexedrine+tDCS+Speech Therapy, Then Placebo+tDCS+Speech Therap
Started | 10
Completed | 10
Not Completed | 0
Period: Washout (1 Week)
Arm/Group | Dexedrine+tDCS+Speech Therapy, Then Placebo+tDCS+Speech Therap
Started | 10
Completed | 10
Not Completed | 0
Period: Placebo+tDCS+Speech Therapy (1 Day)
Arm/Group | Dexedrine+tDCS+Speech Therapy, Then Placebo+tDCS+Speech Therap
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: 10 mg Dexedrine, 1.5 mA anodal tDCS, and speech therapy for 1 day Dexedrine: 10 mg immediate release of Dexedrine Active tDCS: 1.5 mA tDCS anodal tDCS Speech Therapy: 60 min of speech therapy
  Placebo, 1.5 mA anodal tDCS, and speech therapy for 1 day Active tDCS: 1.5 mA tDCS anodal tDCS Speech Therapy: 60 min of speech therapy Placebo
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Non-fluent aphasia assessed by clinicians [Count of Participants; unit: Participants] | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Language Quotient as Assessed by the Western Aphasia Battery
Description: The score on the Language Quotient of the Western Aphasia Battery ranges between 0-100. Higher scores indicate better performance. Below, percent change in the score is reported.
Time Frame: immediately before the treatment, immediately after the treatment
Measure: Mean (95% Confidence Interval); unit: percent change in language quotient
Groups:
- Dexedrine+tDCS+Speech Therapy: The subjects received 10 mg D-AMP 30 minutes before the 60 minutes of SLT; first 20 min is simultaneous tDCS stimulation in this experiment/arm.
- Placebo+tDCS+Speech Therapy: The subjects received placebo 30 minutes before the 60 minutes of SLT; first 20 min is simultaneous tDCS stimulation in this experiment/arm.
Arm/Group | Dexedrine+tDCS+Speech Therapy | Placebo+tDCS+Speech Therapy
Number analyzed (Participants) | 10 | 10
percent change in language quotient | 11.02 [3.22 to 18.81] | -4.2 [-10.57 to 2.26]
Statistical Analysis 1: Comparison: Dexedrine+tDCS+Speech Therapy vs Placebo+tDCS+Speech Therapy; We tested normality using the Kolmogorov-Smirnov (KS) test for all reported measures. We compared scores of Bedside WAB-R® subtests Bedside WAB-R® AQ and LQ from before the study intervention and after the intervention in both experiments by using a two-tailed and paired t-test; Test type: Other — We also performed normalization by calculating the dependent variable as the percentage of change ("proportional change") as it follows; (1) (post-active values - pre-active values)/ (pre-active values) and (2) (post-placebo values - pre-placebo values)/ (pre-placebo series). We compared the percentage of change in Bedside WAB-R® aphasia and language quotients and blood pressures for the experiments with active- and placebo drugs combined active tDCS with MIT using a two-tailed paired t-test; p = 0.008, t-test, 2 sided

2. Primary Outcome: Percent Change in Aphasia Quotient as Assessed by the Western Aphasia Battery
Description: The score on the Aphasia Quotient of the Western Aphasia Battery ranges between 0-100. Higher scores indicate better performance. Below, percent change in the score is reported.
Time Frame: immediately before the treatment, immediately after the treatment
Measure: Mean (95% Confidence Interval); unit: percent change in aphasia quotient
Groups:
- Placebo+tDCS+Speech Therapy: 1.5 mA anodal tDCS, and speech therapy for 1 day
  Active tDCS: 1.5 mA tDCS anodal tDCS
  Speech Therapy: 60 min of speech therapy
  Placebo
Arm/Group | Dexedrine+tDCS+Speech Therapy | Placebo+tDCS+Speech Therapy
Number analyzed (Participants) | 10 | 10
percent change in aphasia quotient | 7.9 [1.49 to 14.31] | -.02 [-7.63 to 7.19]
Statistical Analysis 1: Comparison: Dexedrine+tDCS+Speech Therapy vs Placebo+tDCS+Speech Therapy; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.02, t-test, 2 sided

3. Secondary Outcome: Boston Diagnostic Aphasia Examination
Time Frame: Baseline,2 weeks
Population: Data not collected.
Arm/Group | Dexedrine+tDCS+Speech Therapy | Placebo+tDCS+Speech Therapy
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Boston Diagnostic Aphasia Examination
Time Frame: Baseline,2 months
Population: Data not collected.
Arm/Group | Dexedrine+tDCS+Speech Therapy | Placebo+tDCS+Speech Therapy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percent Change in Blood Pressure
Description: Non-invasive BP measurements performed by a clinician before and after each experiment.
Time Frame: immediately before the treatment, after after the treatment
Measure: Mean (Standard Deviation); unit: percent change in blood pressure
Arm/Group | Dexedrine+tDCS+Speech Therapy | Placebo+tDCS+Speech Therapy
Number analyzed (Participants) | 10 | 10
percent change in blood pressure
  Systolic blood pressure | 10 (3) | 4 (1)
  Diastolic blood pressure | 11 (5) | 5 (2)

ADVERSE EVENTS:
Groups:
- D-AMP+tDCS+Speech Therapy: The subjects received 10 mg of D-AMP medication 30 minutes before the simultaneous tDCS (first 20 min) and 60 min of SLT in this experiment.
- Placebo+tDCS+Speech Therapy: The subjects received placebo medication 30 minutes before the simultaneous tDCS (first 20 min) and 60 min of SLT in this experiment.
Arm/Group | D-AMP+tDCS+Speech Therapy | Placebo+tDCS+Speech Therapy
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/10 | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-AMP+tDCS+Speech Therapy (N=10) | Placebo+tDCS+Speech Therapy (N=10)
Non-significant skin redness and tingling (Skin and subcutaneous tissue disorders) | 9 (9) | 9 (9)
Mild Headache (Nervous system disorders) | 2 (2) | 2 (2) — Resolved shortly after
Mild Insomnia (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The safety phase of the study was completed; however, the efficacy phase was not started.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No